CLINICAL TRIAL: NCT05376813
Title: Elaboration of an Algorithm of Automated Segmentation by Magnetic Resonance Imaging for Bone and Muscles of Shoulder
Brief Title: An Algorithm Creation by Automated Segmentation by MRI for Bone and Muscles of Shoulder
Acronym: SEGMENTATION
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: NO ENROULEMENT
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: APHP220324; 2022-A00301-42 (Registry Identifier: IDRCB)
Record Dates: First submitted 2022-05-09; First posted 2022-05-17 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2024-06

CONDITIONS: Reverse Shoulder Prosthesis
Keywords: Reverse Shoulder Prosthesis; Algorithm; Automatic segmentation; Magnetic resonance imaging; Computed tomography; 3D imaging; Manual segmentation
MeSH Terms: interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Intervention Model Description: No comparative, no control study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental arm (Experimental): All participants are healthy volunteers
  Interventions: Procedure: CT-Scan and MRI

INTERVENTIONS:
Procedure: CT-Scan and MRI — CT-Scan and MRI examination for shoulder will be performed on healthy volunteers.

SUMMARY:
The primary objective of the study is to develop an algorithm of automated segmentation of shoulder by MRI examinations.

DETAILED DESCRIPTION:
This is a national monocentric study which will be conducted in Ambroise Paré hospital of APHP, in orthopaedics department (for enrollment) and radiological department (for CT-scan and MRI examinations) respectively.

Manual segmentations of 5 muscles and 2 bones of shoulder by MRI with automated segmentation of shoulders corresponding to CT-scan imagings.

3D imagings of each shoulder by manual segmentations from MRI and automated segmentation from computed tomography will provide to build a network.

The perspective of the elaborated algorithm should lead to an automated 3D-reconstruction of patients' shoulder as a routine care in surgery.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteer > 18 years, presenting any symptom nor history of shoulder pathology;
* Affiliated to social security scheme.

Exclusion Criteria:

* Symptoms or history of shoulder pathologies;
* Claustrophobia;
* Pregnant woman;
* Patient covered by AME system;
* Contre-indication to perform MRI examination (implant, less 6-months stent implantation, recent surgery, renal insufficiency, pace maker implantation, cardiac defibrillator, cardiovascular catheter, neurostimulation, implantable electronic pompe for automatic injection of medications).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-08-31 (Actual); Primary Completion 2024-04-28 (Actual); Study Completion 2024-04-28 (Actual)

PRIMARY OUTCOMES:
Algorithm developement | through study completion, an average of 8 month
  The developement for automatic segmentation algorithm: uses method with a convolutional neural networks (convolutional neural network - CNN).

CONTACTS AND LOCATIONS:
Overall Officials: Jean-David Werthel, MD, Principal Investigator — Orthopaedics, Ambroise Paré hospital, APHP

IPD SHARING:
Plan to Share IPD: No